CLINICAL TRIAL: NCT03973047
Title: A Phase 1, Randomized Study to Evaluate the Rate of Nausea in Healthy Premenopausal Female Subjects Treated With a Single Dose of Bremelanotide Alone or With Zofran
Brief Title: Study to Evaluate Rate of Nausea in Healthy Premenopausal Female Subjects Treated With Single Dose of Bremelanotide Alone or With Zofran
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMAG-BMT-HSDD-102
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Nausea
Keywords: Nausea; Bremelanotide; BMT; Zofran; ondansetron; premenopausal; healthy women
MeSH Terms: conditions — Nausea | interventions — bremelanotide; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: BMT will be administered in an open-label manner. Administration of Zofran or placebo will be double-blinded using an over-encapsulation (OE) technique . The randomization assignments and code will not be provided to the Sponsor, sites, or subjects until the study database has been locked, except as unblinding is required for non-study personnel in the regulatory reporting of serious adverse events (SAEs) or for other safety-related reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: BMT plus placebo (Placebo Comparator): 1 dose of BMT 1.75 mg via autoinjector plus placebo (dosed 30±5 minutes prior to BMT dosing) on Day 1.
  Interventions: Drug: Bremelanotide; Drug: Placebo
- Group 2: BMT plus Zofran (Active Comparator): 1 dose of BMT 1.75 mg via autoinjector plus Zofran 8 mg (dosed 30±5 minutes prior to BMT dosing) on Day 1.
  Interventions: Drug: Bremelanotide; Drug: Zofran

INTERVENTIONS:
Drug: Bremelanotide — Sterile aqueous solution for injection, provided as an autoinjector pen
  Other Names: BMT
Drug: Zofran — 8 mg tablet (over-encapsulation in a capsule)
  Other Names: ondansetron
  Arms: Group 2: BMT plus Zofran
Drug: Placebo — capsule
  Arms: Group 1: BMT plus placebo

SUMMARY:
This is a Phase 1, randomized study to evaluate the rate of nausea in healthy premenopausal study participants following a single dose of BMT with or without a single 8 mg po dose of Zofran given 30 minutes before BMT dosing.

DETAILED DESCRIPTION:
This is a Phase 1, randomized study to evaluate the rate of nausea in healthy premenopausal study participants following a single dose of BMT with or without a single 8 mg po dose of Zofran given 30 minutes before BMT dosing. The study consists of a 21-day screening period for subject eligibility followed by a 1-day double-blind period in which all subjects receive a single open-label dose of 1.75 mg SC BMT after receiving a single blinded dose of Zofran (ondansetron) 8 mg or placebo. Approximately 228 subjects will be enrolled at up to two study sites in the United States. Safety and tolerability of BMT administration will be summarized and assessed.

ELIGIBILITY:
Key Inclusion Criteria:

1. Willing and able to provide written informed consent prior to participating in the study.
2. Female subjects ≥18 to 55 years of age (inclusive) and premenopausal as defined by the modified STRAW criteria (specifically, Stage -5 [menses variable to regular] through Stage 1 [≥2 skipped cycles and an interval of amenorrhea ≥60 days]).
3. Able to communicate clearly with the Principle Investigator (PI) and staff; able to read English, complete questionnaires, and understand study procedures.
4. Able to complete all screening period evaluations, stay in the clinic testing facility for minimum of 4 hours following dose of BMT.
5. In good general health, free from clinically significant medical or psychiatric illness or disease (as determined by medical/surgical history, physical examination, weight, 12-lead ECG, and clinical laboratory tests).

Key Exclusion Criteria:

1. Postmenopausal female, designated by having amenorrhea for ≥12 months.
2. Has current or recent (within 6 months) history of gastrointestinal disease, or any surgical or medical condition such as Crohn's disease or liver disease, that could potentially alter the absorption, metabolism, or excretion of the study drug.
3. Has any clinically significant medical condition, physical exam finding, or ECG abnormality, or clinically significant abnormal value for hematology, serology, clinical chemistry, or urinalysis at Screening, or at admission to the study center, as assessed by the PI.
4. Has any of the following:

   - History or current diagnosis of uncontrolled hypertension defined as: Two (2) sequential assessments (at least 5 minutes apart and no more than 15 minutes apart) at levels >140 mmHg SBP or 90 mmHg DBP and/or treatment for hypertension that has been changed at least once in the 4 weeks before Screening.

   - Renal dysfunction (creatinine clearance < 80 mL/min using Cockcroft Gault calculation).
5. History or presence of malignancy within the past 5 years, with the exception of adequately treated localized skin cancer (basal cell or squamous cell carcinoma), which is allowed.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 228 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent nausea following BMT with or without concomitant use of Zofran. | 2 Days
  Incidence of treatment-emergent nausea following a single dose of BMT 1.75 mg SC with or without concomitant use of Zofran.

SECONDARY OUTCOMES:
Severity of nausea using a Visual Analog Scale | 2 Days
  "Severity of Nausea Visual Analog Scale", where the range is 0 to 100 and a lower value represents a better outcome
Time to onset of nausea | 2 Days
  The time to onset of nausea
Duration of nausea | 2 Days
  The duration of nausea

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Early Phase Serrvices, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No